CLINICAL TRIAL: NCT05222087
Title: PRIME_LUNG: Primary Radiotherapy In MEtastatic Lung Cancer. A Pilot Study
Brief Title: PRIME_LUNG: Primary Radiotherapy In MEtastatic Lung Cancer - A Pilot Study
Acronym: PRIME_LUNG
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80476
Record Dates: First submitted 2022-01-06; First posted 2022-02-03 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: NSCLC
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: SoC systemic therapy (Active Comparator)
  Interventions: Drug: SoC systemic therapy
- Arm 2: radiotherapy to lung primary, delivered before cycle three of SoC systemic therapy (Experimental)
  Interventions: Radiation: Radiotherapy; Drug: SoC systemic therapy

INTERVENTIONS:
Radiation: Radiotherapy — 35Gy/5# Central 40Gy/5# Large Tumours >5cm (non-central) 36Gy/12# or 40Gy/15# Ultracentral lesions 50Gy/5# Peripheral Tumours ≤5cm
  Arms: Arm 2: radiotherapy to lung primary, delivered before cycle three of SoC systemic therapy
Drug: SoC systemic therapy — Permitted SoC chemoimmunotherapy for squamous patients will include single agent immunotherapy with Pembrolizumab or in combination with Carboplatin or Paclitaxel. Carbo/Paclitaxel/Pembro intravenous infusions are given every 3 weeks for cycle 1-4, followed by ongoing maintainence with Pembrolizumab from Cycle 5. For non-squamous patients, SoC chemoimmunotherapy will include single agent immunotherapy with Pembrolizumab or in combination with Carboplatin or Permetrexed. Carboplatin/Pemetrexed/Pembrolizumab infusions are given every 3 weeks for four cycles followed by maintenance with Pemetrexed/Pembrolizumab from Cycle 5.

SUMMARY:
Outcome for patients diagnosed with advanced lung cancer remains poor; alternative treatment options are urgently needed. Studies in other metastatic cancers indicate radiotherapy to the primary tumour can improve outcomes. The investigators postulate this will also be observed in lung cancer patients. The aim of this pilot study is to assess the safety and feasibility of stereotactic ablative radiotherapy (SABR) to the lung primary prior to standard of care (SoC) systemic therapy in advanced non-small cell lung cancer (NSCLC). Forty patients with advanced (Stage IV) NSCLC will be recruited across the five Peter Mac campuses. Patients will be randomised to receive SoC systemic therapy with or without radiotherapy to the lung primary. Radiotherapy will be delivered before cycle 3 of SoC systemic therapy. Biospecimens will be collected for future translational research. The primary outcome of the study (feasibility of the protocol) will be assessed by the ability to deliver radiotherapy to the lung cancer primary, whilst meeting dose constraints. The study will also 1) evaluate proportion of patients who are willing to be randomised; 2) describe toxicity during the follow up period in each arm; 3) describe progression free survival.

DETAILED DESCRIPTION:
PRIME-Lung is an open-label randomised pilot study designed to assess the safety and feasibility of radiotherapy to the lung primary prior to commencement of standard of care (SOC) systemic therapy in advanced lung cancer. The study is designed to assess the feasibility of the protocol, and will be escalated, without major modification, directly to a randomised phase III design. This will occur if the following objectives are met in ≥ 66% of patients:

1. Receipt of radiotherapy before cycle 3 of systemic therapy.
2. Ability to meet dose constraints in delivering radiotherapy to the lung primary

The secondary objectives are:

* Evaluate proportion of patients who are willing to be randomized.
* To describe toxicity within 90 days of RT delivery
* To describe progression free survival Blood samples for future translational research will also be established.

Newly diagnosed patients with advanced (Stage IV) non-small cell lung cancer (NSCLC) who have received no prior lines of systemic therapy will be invited to participate (refer to protocol for full inclusion/exclusion criteria). Consenting patients will be randomised to either:

* Arm 1: Systemic therapy alone
* Arm 2: Radiotherapy before cycle 3 of systemic therapy

The trial treatment is therefore the addition of radiotherapy before cycle 3 of SOC systemic therapy.

During treatment (standard and experimental arm) participants will be assessed for radiation toxicity and the occurrence of adverse events. The recruitment period is over 18 months, with study visits at Baseline, radiotherapy (patients in Arm 2 only), Cycle 3 of SOC systemic therapy, 12 and 24 weeks after initiation of therapy, and at disease progression. SOC CT Staging scans will occur every 6 weeks from initiation of SOC systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Newly diagnosed, metastatic (stage IV), non-small cell lung cancer (NSCLC), not amenable to curative surgery or curative radiotherapy
* Histological or cytologically documented NSCLC
* EGFR/ALK/ROS1 Wild-type
* Primary disease suitable for radiotherapy and not requiring immediate palliative irradiation
* ECOG 0-1

Exclusion Criteria:

* Medically unfit for systemic therapy
* EGFR/ALK/ROS1 mutation positive
* Has had previous thoracic radiotherapy of > 36Gy in 12 fractions (or equivalent) within the 6 months prior to randomisation.
* Has diagnosed and/or treated additional malignancy within 3 years prior to randomisation with the exception of: curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, curatively treated early-stage cervical cancer, breast cancer or prostate cancer with no evidence of active disease. Other exceptions may be considered following consultation with the principal investigator.
* Has a history of (non-infectious) pneumonitis or current pneumonitis that requires active corticosteroids with a dose equivalent of prednisolone>10mg/d.
* Has had any systemic anti-cancer therapy within 4 weeks prior to randomisation
* A known diagnosis of idiopathic pulmonary fibrosis
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Uncontrolled brain metastases defined as not amenable to surgery or stereotactic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of the study design to be escalated without major modification directly to a randomised phase III design. | 18 months
  To assess the feasibility of the study design to be escalated without major modification directly to a randomised phase III design. Technical feasibility will be assessed by the ability to deliver radiotherapy to the lung cancer primary whilst meeting dose constraints tumour prior to cycle 3 of SoC systemic therapy in metastatic NSCLC.
  Radiotherapy to the primary in stage IV NSCLC will be considered worthwhile to be assessed in a large randomised study if radiotherapy is feasible in >66% of patients randomised to the radiotherapy arm.

SECONDARY OUTCOMES:
willingness to be randomised | 18 months
  evaluate the proportion of patients who are willing to be randomised after being approached for the study.
safety of Radiotherapy addition using NCI CTCAE | 24 months
  The safety of the addition of radiotherapy by describing toxicity during the follow up period in each arm.
  Safety will be measured as adverse events (AE) and serious adverse events (SAEs) using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
PFS | 24 months
  The study will also describe progression free survival within 6 months of follow-up. PFS defined as the time from randomisation to the first occurrence of disease progression, as determined by the Investigator following principles of RECIST 1.1, or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Shankar Siva, A/Prof, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (6):
- Australia (6):
  - Gold Coast University Hospital, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre - Bendigo, Bendigo, Victoria
  - Peter MacCallum Cancer Centre - Monash Cancer Centre, Bentleigh East, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sunshine Hospital Western Health, Sunshine, Victoria

IPD SHARING:
Plan to Share IPD: No